CLINICAL TRIAL: NCT06681389
Title: A Randomized, Double-Blind Phase1b/2a Clinical Study to Evaluate Efficacy, Safety and Tolerability of Subcutaneous Administration of NP-201 Acetate Injection in Healthy Adult Volunteers and in Patients With Mild-To-Moderate Active Ulcerative Colitis
Brief Title: A Study of NP-201 Acetate Injection in Healthy Adult Volunteers and in Patients With Mild-To-Moderate Active Ulcerative Colitis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: NIBEC Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: NIB-IBD-201
Record Dates: First submitted 2024-10-30; First posted 2024-11-08 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Healthy Adult Volunteers; Active Ulcerative Colitis; Active Ulcerative Colitis (UC)
Keywords: Mild-To-Moderate Active Ulcerative Colitis; Ulcerative Colitis; Active Ulcerative Colitis; active ulcerative colitis (UC)
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NP-201 Acetate Injection- Part A (Experimental): 24 healthy participants across 3 cohorts will receive NP-201 acetate injection
  Interventions: Drug: NP-201 acetate injection (Part A)
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NP-201 acetate injection (Part A) — Route of administration- Sub cutaneous. Dosage interval and frequency: MAD1-200mg daily for 5 days; MAD2- 300mg daily for 5 days, MAD3- 400mg daily for 5 days
  Arms: NP-201 Acetate Injection- Part A
Drug: Placebo — Matching placebo administered across Part A and Part B
  Arms: Placebo

SUMMARY:
This Phase 1b/2a clinical development plan is focused on the use of NP-201 acetate injection to investigate the pharmacokinetics (PK), safety, efficacy, PD (pharmacodynamic) markers (Phase 1b) and tolerability of NP-201 acetate injection after subcutaneous (SC) injection of multiple doses in healthy adults and in the ulcerative colitis (UC) patient population.

DETAILED DESCRIPTION:
This Phase 1b/2a randomized, double-blinded study will be conducted in two parts - Phase 1b (Part A) in healthy volunteers and Phase 2a (Part B) in UC patients. This record relates only to Part A/Phase 1b study. This will be updated once Part A is complete.

Part A (Multiple Ascending Doses-MAD): Up to a total of 24 healthy participants will be enrolled into three sequential cohorts (MAD1, MAD2, and MAD3) and randomized 6:2 to receive two dosing regimens of NP-201 acetate injection or placebo daily for 5 days

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females, between 18 to 60 years inclusive, at the time of Screening.
2. Body mass index (BMI) between 18.0 kg/m2 and 32.0 kg/m2(inclusive), at Screening, with a minimum body weight of 50 kg
3. In good health based on the results of medical history, physical examinations, 12-lead ECG, vital signs measurement, and clinical laboratory evaluations at Screening, as assessed by the PI or designee.
4. All female participants of childbearing potential with male sexual partners and male participants with female sexual partners of childbearing potential must consent to use two highly effective methods of contraception from start of study and for at least 90 days (male and female participants) following the EOS visit or last dose of study treatment, whichever is later. Male participants must refrain from sperm donation from start of study and for 90 days after last dose of IP; female participants must refrain from donation of ova from start of study and for 30 days after last dose of IP. WOCBP must have a negative serum pregnancy test at Screening and a negative urine pregnancy test on Screening, and be willing to undergo additional pregnancy tests, as required, throughout the study. Women not of childbearing potential must be postmenopausal (defined as cessation of regular menstrual periods for at least 12 months without an alternative medical cause), confirmed by follicle-stimulating hormone (FSH) level >40 IU/mL at Screening.
5. Participants whose smoking habit in the last 3 months prior to Screening included no more than 14 cigarettes per week (includes e-cigarettes and other nicotine and tobacco products) can be included in the study but must be willing to abstain from smoking from Screening until completion of the EOS visit (Part A only).
6. Ability and willingness to restrict the use of alcohol to ≤ 21 units per week for males and ≤ 14 units per week for females. One unit of alcohol equals ½ pint (285 mL) of beer or lager, 1 glass (125 mL) of wine, or 1/6 gill (25 mL) of spirits. Participants must have negative alcohol breath tests at Screening and Day -1 visits.
7. Participants who are able to receive SC injections specifically participants who have scars or tattoos in the area of concern.
8. Participants must participate voluntarily, sign the ICF, have good compliance, be able and willing to attend the necessary site visits and be willing to cooperate with follow-up visits.
9. No history of severe allergic or anaphylactic reactions, including known allergies or hypersensitivities to NP-201 acetate or its excipients.

Exclusion Criteria:

1. Have a clinically significant medical history or surgical history and have at least one of the following findings:

   1. Have skin diseases that may affect the absorption of the IP (eg, psoriasis, contact dermatitis), scars, tattoos, and skin abnormalities that may interfere with SC injections, or a history of surgery within 60 days of Screening (except for simple appendectomy or hernia repair, as assessed by the PI or designee).
   2. Have a recent significant history of kidney diseases, pancreatitis and/ or nephrolithiasis.
   3. Participants with liver cirrhosis accompanying edema and/or ascites.
   4. Have known clinically significant allergies as assessed by the PI or designee, diseases of either/or the cardiovascular system, peripheral vascular system, skin, mucous membranes, eyes, respiratory system, musculoskeletal system, and/or any other diseases that may pose a problem with the PK evaluation. History of childhood asthma can be included at the discretion of the PI or designee.
   5. Presence of any underlying physical, or psychological medical condition that, in the opinion of the PI or designee, will make it unlikely that the participant will comply with the protocol, or complete the study per the protocol.
2. Pregnant or lactating at Screening or planning to become pregnant at any time during the study, including the follow-up period.
3. Have a clinically relevant history of hypersensitivity reactions or allergic reactions to drugs (such as aspirin and antibiotics), or known drug allergies (eg, to aspirin, nonsteroidal anti-inflammatory drugs [NSAIDs], antibiotics, iodine, anesthetics, other monoclonal antibodies, etc.).
4. Participants who have donated whole blood within 60 days prior to Screening or blood components within 30 days or received blood transfusion within 60 days.
5. Have received an IP or bioequivalence IP in another clinical study or bioequivalence study within 30 days prior to Screening or five half-lives prior to Screening.
6. Use of any prescription drugs within 14 days prior to dosing or non-prescription medications/products, including vitamins, minerals, and phyto-therapeutic/herbal/plant-derived preparations, alternative medicines, or dietary supplements within 7days prior to dosing (at the discretion of the PI or designee). The occasional use of paracetamol(up to 2g/day) is permitted.
7. History of alcoholism, substance or drug abuse-related disorders deemed significant by the PI or designee.
8. Participants with a positive toxicology screening panel. Positive test may be repeated once at the discretion of the investigator.
9. Have positive serology test (hepatitis B surface antigen [HBsAg], or hepatitis C virus antibody [anti-HCV], human immunodeficiency virus [HIV] test,) at Screening.
10. Active infection requiring medical treatment and/or isolation at the time of Screening.
11. Alanine transaminase (ALT), alkaline phosphatase (ALP), aspartate transaminase (AST) > 2.0 × upper limit of normal (ULN).
12. Bilirubin > 1.5 × ULN (isolated bilirubin > 1.5 × ULN is acceptable if bilirubin is fractionated and direct bilirubin < 35%).
13. QTcF > 450 msec for male participants or QTcF > 470 msec for female participants. The QTc is the QT interval corrected for heart rate according to Fridericia's formula (QTcF).
14. Participants with corrected calcium (Ca) > ULN, uric acid > ULN, and/or estimated glomerular filtration rate < 90 mL/min, calculated using Cockroft Gault formula.
15. Others who are ineligible to participate in this clinical study as determined by the PI or designee.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2025-03-25 (Estimated); Study Completion 2025-05-05 (Estimated)

PRIMARY OUTCOMES:
Safety of NP-201 acetate injection in Healthy Volunteers. To evaluate the safety of NP-201 acetate injection by incidence, relationship and severity of adverse events (AE), serious adverse events and Treatment emergent AE | Part A-Screening to Day 12 post first dose administration
Safety of NP-201 acetate injection in Healthy Volunteers. To evaluate the safety of NP-201 acetate injection by changes in baseline Laboratory values | Part A-Screening to Day 12 post first dose administration
Part A-Plasma PK parameters following multiple doses of NP-201 acetate injection- AUC from time 0 to 24 (AUC24) | Part A-Samples collected on Day 1, Day 2, Day 5 and Day 6 post first dose administration
Part A-Plasma PK parameters following multiple doses of NP-201 acetate injection- AUC over the dosing interval (AUCtau) | Part A-Samples collected on Day 1, Day 2, Day 5 and Day 6 post first dose administration
Part A-Plasma PK parameters following multiple doses of NP-201 acetate injection- Area under curve from 0 to last AUC(0-last) | Part A-Samples collected on Day 1, Day 2, Day 5 and Day 6 post first dose administration
Part A-Plasma PK parameters following multiple doses of NP-201 acetate injection- Maximum plasma concentration at steadystate (Cmax,ss) | Part A-Samples collected on Day 1, Day 2, Day 5 and Day 6 post first dose administration
Part A-Plasma PK parameters following multiple doses of NP-201 acetate injection- time to Cmax,ss (tmax,ss) | Part A-Samples collected on Day 1, Day 2, Day 5 and Day 6 post first dose administration
Part A-Plasma PK parameters following multiple doses of NP-201 acetate injection- Apparent oral body clearance at steady-state (CL/Fss) | Part A-Samples collected on Day 1, Day 2, Day 5 and Day 6 post first dose administration
Part A-Plasma PK parameters following multiple doses of NP-201 acetate injection- Apparent volume of distribution at steady-state (Vd/Fss) | Part A- Samples collected on Day 1, Day 2, Day 5 and Day 6 post first dose administration
Part A-Plasma PK parameters following multiple doses of NP-201 acetate injection-Terminal half life (t1/2) | Part A-Samples collected on Day 1, Day 2, Day 5 and Day 6 post first dose administration
Part A-Urine PK parameters of NP-201 acetate injection after multiple doses- cumulative amount of drug excreted in urine (Ae) | Part A-Samples collected on Day 1 and Day 5 post first dose administration
Part A-Urine PK parameters of NP-201 acetate injection after multiple doses- percent fraction of drug recovered in urine (Fe) | Part A-Samples collected on Day 1 and Day 5 post first dose adminstration
Part A-Urine PK parameters of NP-201 acetate injection after multiple doses- Renal clearance (CLr) | Part A-Samples collected on Day 1 and Day 5 post first dose adminstration

SECONDARY OUTCOMES:
Part A- PK of NP-201 acetate injection metabolite- AUC from time 0 to 24 (AUC24) | Part A- Samples collected on Day 1, Day 2, Day 5 and Day 6 post first dose administration
  Plasma Pharmacokinetics in Healthy Volunteers following administration of multiple doses of NP-201 acetate injection by measuring the NP-201 acetate injection metabolite Area under the concentration- time curve from 0 to 24hrs (AUC24)
Part A- PK of NP-201 acetate injection metabolite- AUC over the dosing interval (AUCtau) | Part A- Samples collected on Day 1, Day 2, Day 5 and Day 6 post first dose administration
  Plasma Pharmacokinetics in Healthy Volunteers following administration of multiple doses of NP-201 acetate injection by measuring the NP-201 acetate injection metabolite Area under the concentration- time curve over the dosing interval (AUCtau)
Part A-PK of NP-201 acetate injection metabolite- Maximum plasma concentration at steady state (Cmax,ss) | Part A- Samples collected on Day 1, Day 2, Day 5 and Day 6 post first dose administration
  Plasma Pharmacokinetics in Healthy Volunteers following administration of multiple doses of NP-201 acetate injection by measuring the NP-201 acetate injection metabolite maximum plasma concentration at steady state (CMAX, ss)
Part A- PK of NP-201 acetate Injection metabolite- Time to Cmax,ss (tmax,ss) | Part A- Samples collected on Day 1, Day 2, Day 5 and Day 6 post first dose administration
  Plasma Pharmacokinetics in Healthy Volunteers following administration of multiple doses of NP-201 acetate injection by measuring the NP-201 acetate injection metabolite time to CMAX, ss (tmax, ss)
Part A-PK of NP-201 acetate injection metabolite- Apparent oral body clearance at steady state (CL/Fss) | Part A- Samples collected on Day 1, Day 2, Day 5 and Day 6 post first dose administration
  Plasma Pharmacokinetics in Healthy Volunteers following administration of multiple doses of NP-201 acetate injection by measuring the NP-201 acetate injection metabolite apparent oral body clearance at steady state (CL/Fss)
Part A- PK of NP-201 acetate injection metabolite- Apparent volume of distribution at steady-state (Vd/Fss), | Part A- Samples collected on Day 1, Day 2, Day 5 and Day 6 post first dose administration
  Plasma Pharmacokinetics in Healthy Volunteers following administration of multiple doses of NP-201 acetate injection by measuring the NP-201 acetate injection metabolite apparent volume distribution at steady state (Vd/Fss)
Part A-PK of NP-201 acetate Injection metabolite- terminal half-life (T1/2) | Part A- Samples collected on Day 1, Day 2, Day 5 and Day 6 post first dose administration
  Plasma Pharmacokinetics in Healthy Volunteers following administration of multiple doses of NP-201 acetate injection by measuring the NP-201 acetate injection metabolite terminal half-life (t1/2)

CONTACTS AND LOCATIONS:
Overall Officials: Michele DeSciscio, Dr., Principal Investigator — CMAX Clinical Research Pty Ltd
Locations (1):
- CMAX Clinical Research Pty Ltd, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No